CLINICAL TRIAL: NCT06632171
Title: The Effect of Cognitive Behavioral Therapy-Based and Motivational Interviewing-Supported Psychoeducation on Emotional Eating and Psychological Resilience in Individuals With Obesity
Brief Title: CBT-based and Motivational Interviewing Supported Psychoeducation in Obese Individuals
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Yusuf Durmuş, Lecturer, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Durmusobe
Record Dates: First submitted 2024-10-06; First posted 2024-10-08 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Obesity
Keywords: Obesity, Cognitive Behavioral, Motivational Interviewing
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- psychoeducation 1 (Experimental): Cognitive behavioral therapy- based and motivational interviewing supported psychoeducation will be applied to obese individuals in this group.
  Interventions: Behavioral: Cognitive Behavioral Therapy- Based and Motivational Interviewing-Supported Psychoeducation
- psychoeducation 2 (Experimental): Cognitive behavioral therapy- based and motivational interviewing supported psychoeducation will be applied to obese individuals in this group.
  Interventions: Behavioral: Cognitive Behavioral Therapy- Based and Motivational Interviewing-Supported Psychoeducation
- psychoeducation 3 (Experimental): Cognitive behavioral therapy- based and motivational interviewing supported psychoeducation will be applied to obese individuals in this group.
  Interventions: Behavioral: Cognitive Behavioral Therapy- Based and Motivational Interviewing-Supported Psychoeducation
- psychoeducation 4 (Experimental): Cognitive behavioral therapy- based and motivational interviewing supported psychoeducation will be applied to obese individuals in this group.
  Interventions: Behavioral: Cognitive Behavioral Therapy- Based and Motivational Interviewing-Supported Psychoeducation
- psychoeducation 5 (Experimental): Cognitive behavioral therapy- based and motivational interviewing supported psychoeducation will be applied to obese individuals in this group.
  Interventions: Behavioral: Cognitive Behavioral Therapy- Based and Motivational Interviewing-Supported Psychoeducation
- psychoeducation 6 (Experimental): Cognitive behavioral therapy- based and motivational interviewing supported psychoeducation will be applied to obese individuals in this group.
  Interventions: Behavioral: Cognitive Behavioral Therapy- Based and Motivational Interviewing-Supported Psychoeducation
- psychoeducation 7 (Experimental): Cognitive behavioral therapy- based and motivational interviewing supported psychoeducation will be applied to obese individuals in this group.
  Interventions: Behavioral: Cognitive Behavioral Therapy- Based and Motivational Interviewing-Supported Psychoeducation
- psychoeducation 8 (Experimental): Cognitive behavioral therapy- based and motivational interviewing supported psychoeducation will be applied to obese individuals in this group.
  Interventions: Behavioral: Cognitive Behavioral Therapy- Based and Motivational Interviewing-Supported Psychoeducation
- psychoeducation 9 (Experimental): Cognitive behavioral therapy- based and motivational interviewing supported psychoeducation will be applied to obese individuals in this group.
  Interventions: Behavioral: Cognitive Behavioral Therapy- Based and Motivational Interviewing-Supported Psychoeducation
- psychoeducation 10 (Experimental): Cognitive behavioral therapy- based and motivational interviewing supported psychoeducation will be applied to obese individuals in this group.
  Interventions: Behavioral: Cognitive Behavioral Therapy- Based and Motivational Interviewing-Supported Psychoeducation

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy- Based and Motivational Interviewing-Supported Psychoeducation — The aim of this study is to examine the effects of cognitive-behavioral-based and motivational interview-supported psychoeducation on emotional eating and psychological resilience in obese individuals. The study will be conducted in a randomized controlled experimental design. The sample of the study will consist of 102 obese individuals in total, 51 in the experimental group and 51 in the control group, who meet the inclusion criteria. A cognitive-behavioral and motivational interview-supported psychoeducation program will be applied to the experimental group. All patients will be evaluated at three time points: pretest (baseline), posttest (8 weeks), and follow-up test (3 months after the posttest). No intervention will be applied to the control group.

SUMMARY:
The aim of this study is to examine the effects of cognitive-behavioral and motivational interview-supported psychoeducation on emotional eating and psychological resilience in obese individuals. The study will be conducted with a randomized controlled experimental design. The sample of the study will consist of 102 obese individuals in total, 51 in the experimental group and 51 in the control group, who meet the inclusion criteria. A cognitive-behavioral and motivational interview-supported psychoeducation program will be applied to the experimental group. All patients will be evaluated at three time points: pre-test (baseline), post-test (8 weeks), and follow-up test (3 months after the post-test). No intervention will be applied to the control group. The Emotional Eating Scale and Psychological Resilience Scale will be used as data collection tools in the study. As a result of the study, the hypothesis that the cognitive-behavioral and motivational interview-supported psychoeducation program is effective in reducing the emotional eating levels of obese individuals and increasing their psychological resilience levels will be tested. The findings of the study will contribute to the importance and effectiveness of psychological approaches in the treatment of obesity.

ELIGIBILITY:
Inclusion Criteria:

* Obese individuals (body mass index 30 kg/m2 or more)
* Between the ages of 18-65
* Not having any psychiatric disorder or not using psychiatric medication
* Volunteering to participate in psychoeducation
* Being in a physical and mental condition that will allow them to adapt to treatment
* Signing the informed consent form

Exclusion Criteria:

* Having communication problems
* Having a medical condition (e.g. Cushing syndrome, hypothyroidism) or taking medication that causes obesity
* Having a psychiatric diagnosis (e.g. depression, anxiety disorder, eating disorder) or taking psychotropic medication
* Being pregnant or breastfeeding
* Participating in another diet or exercise program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Emotional eating scale | 2 months
  The lowest score on the scale is "0" and the highest is "30".High scores indicate a bad outcome.
Psychological resilience scale | 2 months
  The lowest score on the scale is "0" and the highest is "84".High scores on the scale indicate a good outcome.